CLINICAL TRIAL: NCT06906744
Title: Quantitative Assessment of Signal Loss in Cardiotocography Using External Recording
Acronym: RCFLoS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9239
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Maternal Heart Rate
Keywords: Maternal heart rate recording; Cardiotocography; Neonatal morbidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Signal loss in cardiotocography (CTG) recordings is numerous and frequent, whether due to artifacts in signal acquisition or confusion over inadvertent maternal heart rate recording, with various negative consequences for neonatal morbidity and unnecessary obstetric interventions. Data on this issue are 10 to 15 years old. CTG remains the primary method for assessing fetal well-being during labor, almost systematically.

ELIGIBILITY:
Inclusion Criteria:

* Adult female (≥ 18 years old)
* Patient treated at a hospital between February 1, 2024 and February 28, 2024
* Having undergone cardiotocography in the labor and delivery room
* Gestational age at delivery >36 weeks

Exclusion Criteria:

* Patient who has expressed opposition to the use of medical record data
* Patient without CTG
* Gestational age at delivery <36 weeks

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Adult female (≥ 18 years old) with gestational age at delivery >36 weeks
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of signal loss during fetal heart rate (FHR) recording during labor. | during labor

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie-Obstétrique CMCO - CHU de Strasbourg - France, Strasbourg, France